CLINICAL TRIAL: NCT03999021
Title: A Phase 1 Open-Label Extension Study to Assess the Long-Term Safety and Tolerability of N-Acetylcysteine (NAC) in Patients With Retinitis Pigmentosa
Brief Title: FIGHT-RP 1 Extension Study
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Zambon SpA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00204017
Record Dates: First submitted 2019-06-24; First posted 2019-06-26 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Retinitis Pigmentosa
MeSH Terms: conditions — Retinitis Pigmentosa

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Experimental Arm (Experimental): All participants to receive study intervention.
  Interventions: Drug: NAC effervescent tablets

INTERVENTIONS:
Drug: NAC effervescent tablets — After completing the pretreatment visits, all patients will enter into the treatment phase where patients will receive 1800 mg of NAC effervescent tablets twice a day. The patients will be followed up every 3 months for 2 years. Therefore, there will be a total of 9 treatment visits (baseline, months 3, 6, 9, 12, 15, 18, 21 and 24).

SUMMARY:
Retinitis Pigmentosa (RP) is a devastating eye disease and at present there are no known treatment options that can alter the rate of vision loss and eventual blindness. In a series of studies in animal models, the effects of exposing cones in the periphery of the retina to a large excess of oxygen results in progressive oxidative damage to cone photoreceptors and cone cell death. Cone cell death gradually spreads from the periphery of the retina toward its center, narrowing the visual field and eventually resulting in tunnel vision. Compared to control patients, those with RP showed significant reduction in the reduced to oxidized glutathione ratio (GSH/GSSG) in aqueous humor and a significant increase in protein carbonyl content. This demonstration of oxidative stress and oxidative damage in the eyes of patients with RP, suggests that oxidative damage-induced cone cell death in animal models of RP may translate to humans with RP and support the hypotheses that (1) potent antioxidants will promote cone survival and function in patients with RP and (2) aqueous GSH/GSSG ratio and carbonyl content on proteins provide useful biomarkers of disease activity in this patient population. Orally administered N-acetylcysteine (NAC) has been found to be a particularly effective antioxidant that promotes prolonged cone survival and maintenance of cone function in a mouse model of RP. Since oral and/or topical administration of NAC is feasible for long-term treatment in humans, and NAC has a good safety profile, there is good rationale to test the effect of NAC in patients with RP.

Oxidative damage has been implicated in several diseases including cystic fibrosis, chronic obstructive pulmonary disease (COPD), and Idiopathic Pulmonary Fibrosis. The effect of oral NAC has been tested in these indications in several clinical trials providing extensive safety data. In COPD, NAC 600mg bid improves airway function and reduces the frequency of acute exacerbations. Doses of up to 1800mg/day have been well-tolerated in the treatment of Idiopathic Pulmonary Fibrosis. Paracetamol (acetaminophen) toxicity is treated with a loading dose of 140 mg/kg NAC followed by 70 mg/kg every 4 hours for 17 doses. Normal volunteers tolerated a dose of 11.2 grams NAC/day for three months without any serious undesirable effects and in another study a dose of 500mg/kg/day was tolerated. The most frequent adverse events associated with the oral administration of NAC are gastrointestinal in nature and include vomiting, diarrhea, stomatitis, abdominal pain and nausea (incidence rate >1/1000 to <1/100). Hypersensitivity reactions including anaphylactic shock and anaphylactic/anaphylactoid reaction (incidence rate <1/10,000), dyspnea, bronchospasm (incidence rate >1/10,000 to <1/1000), angioedema, tachycardia, urticaria, rash and pruritus (incidence rate >1/1000 to <1/100) have been reported less frequently. Finally, reports of headache, tinnitus, pyrexia, blood pressure decreased (incidence rate >1/1000 to <1/100), face edema and hemorrhage have also been collected with oral NAC.

In the FIGHT-RP 1 Study, the investigators used escalating doses of NAC effervescent tablets (from 600 mg in Cohort 1 to 1800 mg in Cohort 3). The maximum tolerated dose was 1800 mg twice a day which will be continued in this study.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years
* Patients diagnosed with RP
* Informed consent
* Authorization of use and disclosure of protected health information

Exclusion Criteria:

* Patients with a concomitant ocular pathology that limits central macular function, including but not limited to: age-related macular degeneration, diabetic retinopathy, and retinal vein occlusion
* Patients with an active ocular infection
* Patients with uncontrolled hypertension (defined as diastolic blood pressure > 95 mm Hg or systolic blood pressure > 160 mm Hg despite medical therapy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-06-24 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Blood Pressure (mmHg) | Up to 2 years
  Blood pressure in mmHg will be used in assessing tolerability of N-Acetylcysteine.
Tolerability of N-Acetylcysteine as assessed by drug-related symptoms | Up to 2 years
  Participants will be assessed for the occurrence of any drug-related symptoms which includes nausea, stomach upset, diarrhea, heartburn, constipation, and vomiting. Based on the number and severity of the symptoms, the physician would conclude whether the patient is tolerating the medication or not.
Tolerability of N-Acetylcysteine as assessed by time at which medication is taken | Up to 2 years
  Medication diary provided to participants will be reviewed to see if participants are taking the medication within the designated time frame.
Tolerability of N-Acetylcysteine as assessed by number of times medication is taken per day | Up to 2 years
  Medication diary provided to participants will be reviewed to see if participants are taking the medication twice a day

SECONDARY OUTCOMES:
Change in best corrected visual acuity (BCVA) | Baseline, every three months up to 2 years
  Scoring is determined by the number of letters gained or lost per month using Early Treatment Diabetic Retinopathy Study (ETDRS) Letter Score and visual acuity score together with an overall score range of 0 to 20/20 where 0 is the worst vision and 20/20 is the best.
Change in central retinal sensitivity as assessed by microperimetry | Baseline, every three months up to 2 years
  Microperimetry (MAIA) is used to test whether there is an increase or decrease in sensitivity (dB) in the retina after initiation of N-Acetylcysteine
Change in ellipsoid zone (EZ) width (µm) | Baseline, every three months up to 2 years
  This will be assessed by spectral domain optical coherence tomography (SD-OCT) after initiation of N-Acetylcysteine.
Change in aqueous reduced to oxidized glutathione ratio (GSH/GSSG) | Baseline, every three months up to 2 years
  This will be calculated from the proportions of reduced glutathione and oxidized glutathione in the aqueous.
Change in serum carbonyl content (nmol/mg) | Baseline, every three months up to 2 years
Change in aqueous levels of N-Acetylcysteine (mg) | Baseline, every 6 months up to 2 years
Change in plasma levels of N-Acetylcysteine (µg/ml) | Baseline, every 3 months up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Peter Campochiaro, Principal Investigator — Johns Hopkins University
Locations (1):
- Wilmer Eye Institute at Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No